CLINICAL TRIAL: NCT05150951
Title: An Attempt at Translating Novelty-enhanced Extinction of Context Conditioning From Rodents to Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-03596
Record Dates: First submitted 2021-11-06; First posted 2021-12-09 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Threat conditioning; Virtual reality; Extinction; Behavioral tagging
MeSH Terms: interventions — Extinction, Biological

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are never told which manipulation that is expected to affect the threat memory processes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Novel exploration is used before extinction in an attempt to strengthen the extinction consolidation.
  Interventions: Behavioral: Novel Exploration; Behavioral: Threat conditioning; Behavioral: Extinction; Behavioral: Reinstatement
- Control group (Experimental): Participants perform a control task (visual attention) instead of the novel exploration.
  Interventions: Behavioral: Threat conditioning; Behavioral: Extinction; Behavioral: Reinstatement; Behavioral: Visual attention control task

INTERVENTIONS:
Behavioral: Novel Exploration — Exploration of a novel 3D-environment in virtual reality.
  Arms: Experimental group
Behavioral: Threat conditioning — Session 1. Threat conditioning to two different (CS+, CS-) virtual reality contexts (i.e rooms). One of these is paired with a mild electric shock. The context paired with the electric shock (CS+) is counterbalanced across participants. Participants are instructed that they may receive electrical shocks during the procedure.
Behavioral: Extinction — Session 2. Participants are repeatedly exposed to the both contexts from session 1 (CS+, CS-), but no shocks are delivered.
Behavioral: Reinstatement — Session 3. Participants are again repeatedly exposed to both contexts from session 1 (CS+, CS-), after a few shocks delivered in a neutral context.
Behavioral: Visual attention control task — Session 2. A visual attention task used as a control task instead of novel exploration.
  Arms: Control group

SUMMARY:
In rodents, novel exploration has been used to strengthen the consolidation of a variety of hippocampal-dependent learning tasks. To our knowledge, no attempt have been made to translate the effect of strengthening the memory of an extinction of a context conditioning memory. This study uses virtual reality for both context conditioning and novel exploration in an attempt at translating these findings from rodents to humans, thus, using novel exploration to strengthen an extinction memory. Threat responses are measured with skin conductance and startle responses. If this effect could be shown experimentally in humans, that experimental setup could become an important tool in understanding important memory processes of fear, such as reconsolidation and behavioral tagging.

DETAILED DESCRIPTION:
The study employs healthy participants and includes three experimental sessions, roughly 24 h apart. During the first session, participants undergo context conditioning in virtual reality where the CS+ and CS- are two different rooms. During the second session, half of the participants perform an exploration of a novel virtual environment, and the other half performs a visual attention task. About 60 min later, participants undergo extinction to the context conditioning performed in session 1, again in virtual reality. In session 3, remaining threat responses are measured through a reinstatement procedure, again in virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and complete study procedures

Exclusion Criteria:

* Current psychiatric disorder.
* Current use of psychotropic medication
* Current use of neurological conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Physiological arousal response during reinstatement. | Day 3
  Startle responses and skin conductance responses are used as measures of physiological arousal response.

SECONDARY OUTCOMES:
Physiological arousal response during extinction | Day 2
  Startle responses and skin conductance responses are used as measures of physiological arousal response
Physiological arousal response during threat conditioning | Day 1
  Startle responses and skin conductance responses are used as measures of physiological arousal response
Subjective fear ratings | Day 1, 2 & 3.
  Subjective ratings of fear (0-100) where 0 is no fear and 100 is worst imaginable fear.
Subjective discomfort ratings | Day 1, 2 & 3
  Subjective ratings of discomfort where 0 is no discomfort and 100 is worst imaginable discomfort.

OTHER OUTCOMES:
Navigation success | Day 2
  Questions designed to probe the amount of navigation performed by participants doing the novel exploration task. Three yes/no question of "Did you find object X?" and then participants are asked to point at their position in a stylized map overviewing the novel exploration context.
State-Trait Anxiety Inventory (STAI-T) | Day 2
  This is a self-rated questionnaire measuring trait anxiety. Higher scores indicate higher level of trait-anxiety (range 20-80).
Generalized anxiety disorder 7 (GAD-7) | Day 2
  This is a self-rated questionnaire for screening and severity measuring of generalized anxiety disorder (range 0-21). Higher scores indicate more symptoms of generalized anxiety.
Patient Health Questionnaire 9 (PHQ-9) | Day 2
  This is a self-rated questionnaire for screening for the presence and severity of depression (0-27). Higher scores indicate a more symptoms, and severity of symptoms, of depression

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ågren, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, deparmtent of Psychology, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymous behavioural data, training material, Statistical Analysis plan, and informed consent form on the project site on Open Science Framework (https://osf.io/4yjev/). Statistical Analysis Plan will be pre-registered on the same site (Open Science Framework).
Supporting Information: SAP, ICF
Time Frame: Data will be available from completion of analysis and publication, and onwards.
Access Criteria: Anonymous behavioural data, training material, Statistical Analysis plan, and informed consent form will be made public on the project site on Open Science Framework (https://osf.io/4yjev/)

REFERENCES:
- [Background] Moncada D, Ballarini F, Viola H. Behavioral Tagging: A Translation of the Synaptic Tagging and Capture Hypothesis. Neural Plast. 2015;2015:650780. doi: 10.1155/2015/650780. Epub 2015 Aug 25. PMID 26380117